CLINICAL TRIAL: NCT01641042
Title: Immunogenicity and Safety Study of GSK Biologicals' Meningococcal Vaccine GSK 134612 Administered to at Risk Subjects From 1 to Less Than 18 Years
Brief Title: Comparison of GlaxoSmithKline (GSK)134612 in Subjects With Increased Risk for Meningococcal Disease Versus Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115524; 2011-002410-36 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-03

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal vaccines; Vaccines, conjugate; Neisseria meningitidis; Immunocompromised patient
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Healthy Group (Experimental): The subjects in the Healthy group will be age-matched to the subjects in the At-risk group. Subjects will receive 2 doses of the investigational vaccine.
  Interventions: Biological: Meningococcal vaccine GSK134612
- At-risk Group (Experimental): This group includes subjects with medical conditions placing them at an increased risk for meningococcal disease. Subjects will receive 2 doses of the investigational vaccine.
  Interventions: Biological: Meningococcal vaccine GSK134612

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — 2 doses of the vaccine administered intramuscularly in the anterolateral thigh muscle of the non-dominant leg for subjects aged 12 months to 2 years and in the deltoid of the non-dominant arm for older subjects.

SUMMARY:
The purpose of this study is to investigate the immunogenicity, reactogenicity and safety of the new meningococcal vaccine 134612 in subjects with increased risk of meningococcal disease and compare it to its activity in healthy subjects.

DETAILED DESCRIPTION:
For each at risk subject enrolled, an age-matched healthy subject will be enrolled. Age matching will be performed according to the following age strata: 1-5 years, 6-10 years, 11-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* A male or female 1 to 17 years of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject and informed assent obtained from the subject, if appropriate, prior to enrolment.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if

  * the subject has practiced adequate contraception for one month (30 days) prior to the first vaccine dose, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception from administration of the first vaccine dose until 2 months after administration of the second vaccine dose.

Additional inclusion criterion for At-risk group • Subjects with an increased risk for meningococcal disease, such as anatomic asplenia or some degree of functional asplenia or complement deficiencies.

Additional inclusion criteria for Healthy group

* Healthy subject as established by medical history and clinical examination before entering into the study.
* Age-matched to a subject from the At-risk group according to age strata 1-5 years, 6-10 years and 11 to 17 years.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period (until the phone contact at Month 8).
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting 30 days before administration of each study vaccine dose until 30 days after administration of each study vaccine dose. Administration of licensed inactivated influenza vaccines is allowed as per local recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of meningococcal disease.
* Any confirmed or suspected Human Immunodeficiency Virus (HIV) infection, based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine until one month after the second dose of study vaccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine including latex.
* Major congenital defects.
* History of any neurological disorders or seizures, including Guillain-Barré syndrome (GBS). History of a simple, single febrile seizure is permitted.
* Acute disease and/or fever at the time of enrolment.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Additional exclusion criteria for the At-risk group

• Vaccination against meningococcal disease of any serogroup

* within the last 3 years for subjects younger than 7 years.
* within the last 5 years for subjects 7 years and older.

Additional exclusion criteria for the Healthy group

* Vaccination against meningococcal disease of any serogroup with polysaccharide or conjugate vaccine within the last 5 years.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* Serious chronic illness.
* History of asplenia or hyposplenia or complement deficiencies.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2012-09-10; Primary Completion 2014-10-10 (Actual); Study Completion 2015-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (12):
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Durham, North Carolina
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix At-Risk Group: Male or female subjects, aged 1 to 17 years of age, with an increased risk for meningococcal disease due to anatomic asplenia or some degree of functional asplenia, who received 2 doses of the Nimenrix vaccine at Month 0 and Month 2. The vaccine was administered intramuscularly in the anterolateral thigh muscle of the non-dominant leg for subjects aged 12 months to 2 years and in the deltoid of the non-dominant arm for older subjects.
- Nimenrix Healthy Group: Healthy male or female subjects, aged 1 to 17 years of age, who received 2 doses of the Nimenrix vaccine at Month 0 and Month 2, administered intramuscularly in the anterolateral thigh muscle of the non-dominant leg for subjects aged 12 months to 2 years and in the deltoid of the non-dominant arm for older subjects.
Period: Overall Study
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Started | 43 | 43
Completed | 43 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.0 (4.4) | 11.5 (3.6) | 11.75 (4.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 23 | 21 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/African American | 11 | 2 | 13
  American Indian or Alaskan Native | 0 | 2 | 2
  White-Caucasian/European Heritage | 32 | 38 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Vaccine Response for Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitides Serogroups A, C, W-135 and Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY) Antibodies
Description: Vaccine response was defined as: rSBA antibody titers greater than or equal to (≥) 1:32, for initially seronegative subjects [i.e. pre-vaccination rSBA antibody titers below (<) 1:8] and at least a 4-fold increase in rSBA antibody titers from pre to post-vaccination, for initially seropositive subjects (i.e. pre-vaccination rSBA antibody titers ≥ 1:8).
Time Frame: One month after the first vaccine dose (at Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all eligible subjects who complied with the blood sample schedule for Visit 2 (Month 1) and Visit 4 (Month 3), for whom data concerning immunogenicity endpoint measures were available for at least one antigen component of the vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Participants
  rSBA-MenA | 40 | 39
  rSBA-MenC | 37 | 39
  rSBA-MenW-135 | 40 | 39
  rSBA-MenY | 39 | 40

2. Primary Outcome: Number of Subjects With a Vaccine Response for Serum Bactericidal Assay Using Human Complement Against N. Meningitides Serogroups A, C, W-135 and Y (hSBA-MenA, hSBA-MenC, hSBA-MenW-135, hSBA-MenY) Antibodies
Description: Vaccine response was defined as: hSBA antibody titers ≥ 1:8, for initially seronegative subjects (i.e. pre-vaccination rSBA antibody titers < 1:4) and at least a 4-fold increase in hSBA antibody titers from pre to post-vaccination, for initially seropositive subjects (i.e. pre-vaccination rSBA antibody titers ≥ 1:4).
Time Frame: One month after the first vaccine dose (at Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all eligible subjects who complied with the blood sample schedule for Visit 2 (Month 1) and Visit 4 (Month 3), for whom data concerning immunogenicity endpoint measures were available for at least one antigen component of the vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 38 | 38
Participants
  hSBA-MenA: number analyzed (Participants) | 33 | 33
  hSBA-MenA | 23 | 23
  hSBA-MenC: number analyzed (Participants) | 35 | 33
  hSBA-MenC | 27 | 20
  hSBA-MenW-135: number analyzed (Participants) | 36 | 32
  hSBA-MenW-135 | 20 | 21
  hSBA-MenY | 23 | 29

3. Secondary Outcome: Number of Subjects With a Vaccine Response for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibodies
Description: Vaccine response was defined as: rSBA antibody titers ≥ 1:32, for initially seronegative subjects (i.e. pre-vaccination rSBA antibody titers < 1:8) and at least a 4-fold increase in rSBA antibody titers from pre to post-vaccination, for initially seropositive subjects (i.e. pre-vaccination rSBA antibody titers ≥ 1:8).
Time Frame: One month after the second vaccine dose (At Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 39 | 39
Participants
  rSBA-MenA | 39 | 39
  rSBA-MenC | 39 | 39
  rSBA-MenW-135 | 39 | 39
  rSBA-MenY | 39 | 39

4. Secondary Outcome: Number of Subjects With a Vaccine Response to hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibodies
Description: as for outcome 2
Time Frame: One month after the second vaccine dose (At Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 37 | 37
Participants
  hSBA-MenA: number analyzed (Participants) | 33 | 32
  hSBA-MenA | 28 | 24
  hSBA-MenC: number analyzed (Participants) | 34 | 34
  hSBA-MenC | 34 | 29
  hSBA-MenW-135: number analyzed (Participants) | 36 | 31
  hSBA-MenW-135 | 29 | 24
  hSBA-MenY | 27 | 27

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off value for the assay was ≥ 1:8.
Time Frame: At pre-primary vaccination (Month 0), at post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Participants
  rSBA-MenA; Month 0 | 7 | 2
  rSBA-MenA; Month 1 | 40 | 40
  rSBA-MenA; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenA; Month 3 | 39 | 39
  rSBA-MenC; Month 0 | 10 | 5
  rSBA-MenC; Month 1 | 37 | 39
  rSBA-MenC; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenC; Month 3 | 39 | 39
  rSBA-MenW-135; Month 0 | 5 | 3
  rSBA-MenW-135; Month 1 | 40 | 39
  rSBA-MenW-135; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenW-135; Month 3 | 39 | 39
  rSBA-MenY; Month 0 | 9 | 8
  rSBA-MenY; Month 1 | 40 | 40
  rSBA-MenY; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenY; Month 3 | 39 | 39

6. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off value for the assay was ≥ 1:128.
Time Frame: Pre-primary vaccination at Month 0, post first vaccine dose at Month 1 and post second vaccine dose at Month 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Participants
  rSBA-MenA; Month 0 | 6 | 1
  rSBA-MenA; Month 1 | 40 | 40
  rSBA-MenA; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenA; Month 3 | 39 | 39
  rSBA-MenC; Month 0 | 3 | 4
  rSBA-MenC; Month 1 | 37 | 39
  rSBA-MenC; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenC; Month 3 | 38 | 38
  rSBA-MenW-135; Month 0 | 4 | 2
  rSBA-MenW-135; Month 1 | 40 | 39
  rSBA-MenW-135; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenW-135; Month 3 | 38 | 39
  rSBA-MenY; Month 0 | 8 | 8
  rSBA-MenY; Month 1 | 40 | 40
  rSBA-MenY; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenY; Month 3 | 39 | 39

7. Secondary Outcome: Antibody Titers for rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY Meningococcal Antigens
Description: Antibody titers were measured in geometric mean titers (GMTs), calculated on all subjects.
Time Frame: At pre-primary vaccination (Month 0), post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Titers
  rSBA-MenA; Month 0 | 8.6 [4.8 to 15.3] | 4.8 [3.6 to 6.3]
  rSBA-MenA; Month 1 | 2012.8 [1414 to 2865.3] | 4025.6 [3065.1 to 5287.2]
  rSBA-MenA; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenA; Month 3 | 2820.1 [1899 to 4187.9] | 3553.1 [2640.3 to 4781.5]
  rSBA-MenC; Month 0 | 9 [5.4 to 15] | 6.3 [4.2 to 9.3]
  rSBA-MenC; Month 1 | 1374.8 [693.4 to 2725.7] | 2233.4 [1197.4 to 4165.6]
  rSBA-MenC; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenC; Month 3 | 1684.3 [1097.8 to 2584.1] | 1684.3 [1087.8 to 2608.1]
  rSBA-MenW-135; Month 0 | 7 [4.2 to 11.7] | 5.1 [3.8 to 6.9]
  rSBA-MenW-135; Month 1 | 3050.9 [2029.8 to 4585.5] | 4167.6 [2620 to 6629.2]
  rSBA-MenW-135; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenW-135; Month 3 | 5844.3 [4046.3 to 8441.3] | 6981.1 [5467.9 to 8913]
  rSBA-MenY; Month 0 | 10.6 [5.7 to 19.7] | 9.7 [5.4 to 17.3]
  rSBA-MenY; Month 1 | 4624.2 [3125.5 to 6841.6] | 7009 [5175.6 to 9491.9]
  rSBA-MenY; Month 3: number analyzed (Participants) | 39 | 39
  rSBA-MenY; Month 3 | 5640.2 [4142.5 to 7679.5] | 6618.6 [4875.6 to 8984.6]

8. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBAMenW-135 and hSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off value for the assay was ≥ 1:4.
Time Frame: Pre-primary vaccinarion (Month 0), post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Participants
  hSBA-MenA; Month 0: number analyzed (Participants) | 36 | 35
  hSBA-MenA; Month 0 | 14 | 12
  hSBA-MenA; Month 1: number analyzed (Participants) | 35 | 37
  hSBA-MenA; Month 1 | 29 | 28
  hSBA-MenA; Month 3: number analyzed (Participants) | 37 | 36
  hSBA-MenA; Month 3 | 35 | 29
  hSBA-MenC; Month 0: number analyzed (Participants) | 36 | 35
  hSBA-MenC; Month 0 | 21 | 23
  hSBA-MenC; Month 1: number analyzed (Participants) | 37 | 38
  hSBA-MenC; Month 1 | 34 | 36
  hSBA-MenC; Month 3: number analyzed (Participants) | 38 | 39
  hSBA-MenC; Month 3 | 38 | 39
  hSBA-MenW-135; Month 0: number analyzed (Participants) | 37 | 33
  hSBA-MenW-135; Month 0 | 20 | 16
  hSBA-MenW-135; Month 1: number analyzed (Participants) | 37 | 39
  hSBA-MenW-135; Month 1 | 34 | 39
  hSBA-MenW-135; Month 3: number analyzed (Participants) | 39 | 38
  hSBA-MenW-135; Month 3 | 39 | 38
  hSBA-MenY; Month 0: number analyzed (Participants) | 38 | 38
  hSBA-MenY; Month 0 | 24 | 25
  hSBA-MenY; Month 1 | 37 | 40
  hSBA-MenY; Month 3: number analyzed (Participants) | 39 | 39
  hSBA-MenY; Month 3 | 39 | 39

9. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBAMenW-135 and hSBA-MenY Titers ≥ the Cut-off Values
Description: The cut-off value for the assay ≥ 1:8.
Time Frame: Pre-primary vaccinarion (Month 0), post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Participants
  hSBA-MenA; Month 0: number analyzed (Participants) | 36 | 35
  hSBA-MenA; Month 0 | 13 | 12
  hSBA-MenA; Month 1: number analyzed (Participants) | 35 | 37
  hSBA-MenA; Month 1 | 29 | 28
  hSBA-MenA; Month 3: number analyzed (Participants) | 37 | 36
  hSBA-MenA; Month 3 | 35 | 29
  hSBA-MenC; Month 0: number analyzed (Participants) | 36 | 35
  hSBA-MenC; Month 0 | 20 | 22
  hSBA-MenC; Month 1: number analyzed (Participants) | 37 | 38
  hSBA-MenC; Month 1 | 34 | 36
  hSBA-MenC; Month 3: number analyzed (Participants) | 38 | 39
  hSBA-MenC; Month 3 | 38 | 39
  hSBA-MenW-135; Month 0: number analyzed (Participants) | 37 | 33
  hSBA-MenW-135; Month 0 | 20 | 16
  hSBA-MenW-135; Month 1: number analyzed (Participants) | 37 | 39
  hSBA-MenW-135; Month 1 | 34 | 39
  hSBA-MenW-135; Month 3: number analyzed (Participants) | 39 | 38
  hSBA-MenW-135; Month 3 | 39 | 38
  hSBA-MenY; Month 0: number analyzed (Participants) | 38 | 38
  hSBA-MenY; Month 0 | 24 | 25
  hSBA-MenY; Month 1 | 37 | 40
  hSBA-MenY; Month 3: number analyzed (Participants) | 39 | 39
  hSBA-MenY; Month 3 | 39 | 39

10. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Meningococcal Antigens
Description: Antibody titers were measured in Geometric mean titers (GMTs), calculated on all subjects.
Time Frame: Pre-primary vaccination at Month 0, post first vaccine dose at Month 1 and post second vaccine dose at Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 40
Titres
  hSBA-MenA; Month 0: number analyzed (Participants) | 36 | 35
  hSBA-MenA; Month 0 | 5.5 [3.4 to 8.9] | 4.2 [2.9 to 6.1]
  hSBA-MenA; Month 1: number analyzed (Participants) | 35 | 37
  hSBA-MenA; Month 1 | 105.9 [47.6 to 235.6] | 68.7 [32.6 to 144.5]
  hSBA-MenA; Month 3: number analyzed (Participants) | 37 | 36
  hSBA-MenA; Month 3 | 235.1 [136.2 to 405.9] | 90.3 [44.8 to 182.1]
  hSBA-MenC; Month 0: number analyzed (Participants) | 36 | 35
  hSBA-MenC; Month 0 | 12.9 [6.5 to 25.7] | 10.9 [6.3 to 18.6]
  hSBA-MenC; Month 1: number analyzed (Participants) | 37 | 38
  hSBA-MenC; Month 1 | 812.9 [283.5 to 2330.9] | 196.7 [84.6 to 457.2]
  hSBA-MenC; Month 3: number analyzed (Participants) | 38 | 39
  hSBA-MenC; Month 3 | 1472.1 [733.6 to 2954] | 764.6 [404.8 to 1444.5]
  hSBA-MenW-135; Month 0: number analyzed (Participants) | 37 | 33
  hSBA-MenW-135; Month 0 | 21.7 [9.9 to 47.7] | 13.6 [6.4 to 28.5]
  hSBA-MenW-135; Month 1: number analyzed (Participants) | 37 | 39
  hSBA-MenW-135; Month 1 | 283.7 [137.4 to 585.6] | 263.7 [187.3 to 371.2]
  hSBA-MenW-135; Month 3: number analyzed (Participants) | 39 | 38
  hSBA-MenW-135; Month 3 | 884.5 [567.2 to 1379.2] | 590.8 [443 to 787.8]
  hSBA-MenY; Month 0: number analyzed (Participants) | 38 | 38
  hSBA-MenY; Month 0 | 37 [16.7 to 82.4] | 32 [15.5 to 65.8]
  hSBA-MenY; Month 1 | 743.6 [352.9 to 1566.7] | 661.7 [460.2 to 951.6]
  hSBA-MenY; Month 3: number analyzed (Participants) | 39 | 39
  hSBA-MenY; Month 3 | 1415.1 [905.2 to 2212.2] | 800.7 [638.1 to 1004.7]

11. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations ≥ the Cut-off Values
Description: The cut-off value for the assay was ≥ 0.3 micrograms per milliliter (μg/m).
Time Frame: Pre-primary vaccinarion (Month 0), post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 33 | 34
Participants
  anti-PSA; Month 0: number analyzed (Participants) | 28 | 30
  anti-PSA; Month 0 | 28 | 30
  anti-PSA; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSA; Month 1 | 29 | 34
  anti-PSA; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSA; Month 3 | 33 | 32
  anti-PSC; Month 0 | 15 | 4
  anti-PSC; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSC; Month 1 | 29 | 34
  anti-PSC; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSC; Month 3 | 33 | 32
  anti-PSW-135; Month 0: number analyzed (Participants) | 28 | 30
  anti-PSW-135; Month 0 | 21 | 19
  anti-PSW-135; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSW-135; Month 1 | 29 | 34
  anti-PSW-135; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSW-135; Month 3 | 33 | 32
  anti-PSY; Month 0: number analyzed (Participants) | 7 | 5
  anti-PSY; Month 0 | 7 | 5
  anti-PSY; Month 1: number analyzed (Participants) | 10 | 13
  anti-PSY; Month 1 | 10 | 13
  anti-PSY; Month 3: number analyzed (Participants) | 10 | 11
  anti-PSY; Month 3 | 10 | 11

12. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentration ≥ the Cut-off Values
Description: The cut-off value for the assay was ≥ 2.0 μg/mL.
Time Frame: Pre-primary vaccinarion (Month 0), post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 33 | 34
Participants
  anti-PSA; Month 0: number analyzed (Participants) | 28 | 30
  anti-PSA; Month 0 | 12 | 9
  anti-PSA; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSA; Month 1 | 29 | 34
  anti-PSA; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSA; Month 3 | 33 | 32
  anti-PSC; Month 0 | 3 | 2
  anti-PSC; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSC; Month 1 | 26 | 32
  anti-PSC; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSC; Month 3 | 30 | 27
  anti-PSW-135; Month 0: number analyzed (Participants) | 28 | 30
  anti-PSW-135; Month 0 | 4 | 2
  anti-PSW-135; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSW-135; Month 1 | 28 | 33
  anti-PSW-135; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSW-135; Month 3 | 33 | 32
  anti-PSY; Month 0: number analyzed (Participants) | 7 | 5
  anti-PSY; Month 0 | 3 | 3
  anti-PSY; Month 1: number analyzed (Participants) | 10 | 13
  anti-PSY; Month 1 | 10 | 13
  anti-PSY; Month 3: number analyzed (Participants) | 10 | 11
  anti-PSY; Month 3 | 10 | 11

13. Secondary Outcome: Antibody Titers for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Meningococcal Antigens
Description: Antibody titers were measured in geometric mean concentrations (GMCs), calculated on all subjects.
Time Frame: Pre-primary vaccinarion (Month 0), post first vaccine dose (Month 1) and post second vaccine dose (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 33 | 34
Titers
  anti-PSA; Month 0: number analyzed (Participants) | 28 | 30
  anti-PSA; Month 0 | 1.9 [1.5 to 2.4] | 1.4 [1.1 to 1.8]
  anti-PSA; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSA; Month 1 | 17.4 [11.7 to 25.8] | 16.2 [11.3 to 23.3]
  anti-PSA; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSA; Month 3 | 14.2 [10.5 to 19.3] | 10.7 [8 to 14.3]
  anti-PSC; Month 0 | 0.4 [0.2 to 0.6] | 0.2 [0.1 to 0.3]
  anti-PSC; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSC; Month 1 | 8.3 [5.6 to 12.5] | 8.4 [5.9 to 11.8]
  anti-PSC; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSC; Month 3 | 6 [4.4 to 8.1] | 5.8 [4.2 to 8]
  anti-PSW-135; Month 0: number analyzed (Participants) | 28 | 30
  anti-PSW-135; Month 0 | 0.6 [0.3 to 1.1] | 0.4 [0.3 to 0.6]
  anti-PSW-135; Month 1: number analyzed (Participants) | 29 | 34
  anti-PSW-135; Month 1 | 14.9 [8.4 to 26.3] | 13.3 [9.2 to 19.4]
  anti-PSW-135; Month 3: number analyzed (Participants) | 33 | 32
  anti-PSW-135; Month 3 | 19 [12.8 to 28.2] | 14 [9.9 to 19.8]
  anti-PSY; Month 0: number analyzed (Participants) | 7 | 5
  anti-PSY; Month 0 | 2.9 [1.1 to 7.9] | 2.5 [1 to 6.1]
  anti-PSY; Month 1: number analyzed (Participants) | 10 | 13
  anti-PSY; Month 1 | 20.4 [6.3 to 66.2] | 17.3 [11.2 to 26.8]
  anti-PSY; Month 3: number analyzed (Participants) | 10 | 11
  anti-PSY; Month 3 | 30 [10.4 to 86.5] | 12.5 [9.4 to 16.7]

14. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms at Age Stratum 1-5 Years
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented and with their symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 3 | 3
Participants
  Any Pain, Dose 1 | 2 | 0
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 2 | 0
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 2 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 3 | 2
  Any Pain, Dose 2 | 1 | 1
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Pain, Dose 2 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 3 | 2
  Any Redness, Dose 2 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 3 | 2
  Any Swelling, Dose 2 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Across Doses | 2 | 1
  Grade 3 Pain, Across Doses | 0 | 0
  Any Redness, Across Doses | 2 | 0
  Grade 3 Redness, Across Doses | 0 | 0
  Any Swelling, Across Doses | 2 | 0
  Grade 3 Swelling, Across Doses | 0 | 0

15. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms at Age Stratum 6-17 Years
Description: Assessed solicited local symptoms were pain, redness and swelling. Any was defined as occurrence of the symptom regardless of intensity grade. Grade 3 pain was defined as cried when limb was moved/spontaneously painful. Grade 3 redness/swelling was defined as redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 39
Participants
  Any Pain, Dose 1 | 28 | 23
  Grade 3 Pain, Dose 1 | 2 | 1
  Any Redness, Dose 1 | 7 | 13
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 12 | 8
  Grade 3 Swelling, Dose 1 | 2 | 2
  Any Pain, Dose 2: number analyzed (Participants) | 38 | 38
  Any Pain, Dose 2 | 29 | 24
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Pain, Dose 2 | 3 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 38 | 38
  Any Redness, Dose 2 | 12 | 8
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 38 | 38
  Any Swelling, Dose 2 | 12 | 10
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Swelling, Dose 2 | 3 | 2
  Any Pain, Across Doses | 32 | 28
  Grade 3 Pain, Across Doses | 4 | 2
  Any Redness, Across Doses | 14 | 14
  Grade 3 Redness, Across Doses | 1 | 0
  Any Swelling, Across Doses | 18 | 12
  Grade 3 Swelling, Across Doses | 4 | 3

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms at Age Stratum 1-5 Years
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptoms = symptoms which prevented normal everyday activities. Grade 3 fever = oral temperature >39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 3 | 3
Participants
  Any Drowsiness, Dose 1 | 3 | 1
  Grade 3 Drowsiness, Dose 1 | 1 | 0
  Related Drowsiness, Dose 1 | 3 | 0
  Any Irritability, Dose 1 | 2 | 1
  Grade 3 Irritability, Dose 1 | 1 | 0
  Related Irritability, Dose 1 | 2 | 0
  Any Loss of appetite, Dose 1 | 2 | 0
  Grade 3 Loss of appetite, Dose 1 | 0 | 0
  Related Loss of appetite, Dose 1 | 2 | 0
  Any Fever, Dose 1 | 0 | 0
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 0 | 0
  Any Drowsiness, Dose 2: number analyzed (Participants) | 3 | 2
  Any Drowsiness, Dose 2 | 0 | 1
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Drowsiness, Dose 2 | 0 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 3 | 2
  Related Drowsiness, Dose 2 | 0 | 1
  Any Irritability, Dose 2: number analyzed (Participants) | 3 | 2
  Any Irritability, Dose 2 | 0 | 1
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Irritability, Dose 2 | 0 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 3 | 2
  Related Irritability, Dose 2 | 0 | 1
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 3 | 2
  Any Loss of appetite, Dose 2 | 0 | 0
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Loss of appetite, Dose 2 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 3 | 2
  Related Loss of appetite, Dose 2 | 0 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 3 | 2
  Any Fever, Dose 2 | 0 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 3 | 2
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 3 | 2
  Related Fever, Dose 2 | 0 | 0
  Any Drowsiness, Across doses | 3 | 2
  Grade 3 Drowsiness, Across doses | 1 | 0
  Related Drowsiness, Across doses | 3 | 1
  Any Irritability, Across doses | 2 | 2
  Grade 3 Irritability, Across doses | 1 | 0
  Related Irritability, Across doses | 2 | 1
  Any Loss of appetite, Across doses | 2 | 0
  Grade 3 Loss of appetite, Across doses | 0 | 0
  Related Loss of appetite, Across doses | 2 | 0
  Any Fever, Across doses | 0 | 0
  Grade 3 Fever, Across doses | 0 | 0
  Related Fever, Across doses | 0 | 0

17. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms at Age Stratum 6-17 Years
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache and fever. Gastrointestinal symptoms include nausea, vomiting, diarrhoea and/or abdominal pain. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptoms = symptoms which prevented normal everyday activities. Grade 3 fever = oral temperature >39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 40 | 39
Participants
  Any Fatigue, Dose 1 | 18 | 12
  Grade 3 Fatigue, Dose 1 | 1 | 0
  Related Fatigue, Dose 1 | 17 | 12
  Any Gastrointestinal, Dose 1 | 5 | 3
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0
  Related Gastrointestinal, Dose 1 | 4 | 3
  Any Headache, Dose 1 | 12 | 9
  Grade 3 Headache, Dose 1 | 0 | 0
  Related Headache, Dose 1 | 9 | 9
  Any Fever, Dose 1 | 3 | 0
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 2 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 38 | 38
  Any Fatigue, Dose 2 | 13 | 7
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Fatigue, Dose 2 | 0 | 1
  Related Fatigue, Dose 2: number analyzed (Participants) | 38 | 38
  Related Fatigue, Dose 2 | 13 | 6
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 38 | 38
  Any Gastrointestinal, Dose 2 | 1 | 6
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Gastrointestinal, Dose 2 | 0 | 2
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 38 | 38
  Related Gastrointestinal, Dose 2 | 1 | 3
  Any Headache, Dose 2: number analyzed (Participants) | 38 | 38
  Any Headache, Dose 2 | 7 | 5
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Headache, Dose 2 | 0 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 38 | 38
  Related Headache, Dose 2 | 6 | 4
  Any Fever, Dose 2: number analyzed (Participants) | 38 | 38
  Any Fever, Dose 2 | 1 | 2
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 38 | 38
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 38 | 38
  Related Fever, Dose 2 | 1 | 1
  Any Fatigue, Across doses | 21 | 14
  Grade 3 Fatigue, Across doses | 1 | 1
  Related Fatigue, Across doses | 21 | 14
  Any Gastrointestinal, Across doses | 6 | 8
  Grade 3 Gastrointestinal, Across doses | 0 | 2
  Related Gastrointestinal, Across doses | 5 | 5
  Any Headache, Across doses | 16 | 10
  Grade 3 Headache, Across doses | 0 | 1
  Related Headache, Across doses | 14 | 10
  Any Fever, Across doses | 4 | 2
  Grade 3 Fever, Across doses | 0 | 0
  Related Fever, Across doses | 3 | 1

18. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type 1 diabetes and allergies.
Time Frame: From Month 0 until the end of the Extended Safety Follow-Up [ESFU] (at Month 8)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

19. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event (AE) covers any untoward medical occurrence in a clinical subject investigation temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an AE reported in addition to those solicited during the clinical study. Also any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE.
Time Frame: During the 31-day (Days 0-30) post first vaccination period
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 43 | 43
Participants | 7 | 7

20. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical subject investigation temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an AE reported in addition to those solicited during the clinical study. Also any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE.
Time Frame: During the 31-day (Days 0-30) post second vaccination period
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 43 | 43
Participants | 3 | 8

21. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 until the end of the ESFU (at Month 8)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix At-Risk Group | Nimenrix Healthy Group
Number analyzed (Participants) | 43 | 43
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period, Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period; SAEs: from Month 0 up to the end of the ESFU Phase (at Month 8).
Arm/Group | Nimenrix At-risk Group | Nimenrix Healthy Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 4/43 | 1/43
Other Adverse Events (participants affected / at risk) | 38/43 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix At-risk Group (N=43) | Nimenrix Healthy Group (N=43)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cystitis escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix At-risk Group (N=43) | Nimenrix Healthy Group (N=43)
Erythema (Skin and subcutaneous tissue disorders) | 16 (21) | 14 (21)
Fatigue (General disorders) | 21 (31) | 14 (19)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (6) | 8 (9)
Headache (Nervous system disorders) | 16 (19) | 10 (14)
Pain (General disorders) | 34 (60) | 29 (48)
Pyrexia (General disorders) | 5 (5) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Swelling (General disorders) | 20 (26) | 12 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.